CLINICAL TRIAL: NCT03616847
Title: Evaluation of Post-operative Swelling and Functional Outcomes in Relation to Pneumatic Tourniquet Use Pattern in Bunion Surgery
Brief Title: Comparison of Different Tourniquet Release Times in Bunion Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Golden Jubilee National Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18/ORTH/03
Record Dates: First submitted 2018-07-25; First posted 2018-08-06 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Hallux Valgus; Hallux Rigidus
Keywords: Randomised controlled trial; Hallux valgus correction; Hallux rigidus correction; Tourniquet; Foot volume
MeSH Terms: conditions — Hallux Valgus; Hallux Rigidus | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Two randomised study groups with one having standard care and the other the intervention.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Those collecting and analysis the data will be masked to the treatment groups. It is not possible to mask the participant or the care provider in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (Experimental): Participants will have hallux valgus/hallux rigidus surgery using a calf tourniquet which will remain inflated until the wound is closed.
  Interventions: Other: Standard care
- Tourniquet release (Experimental): Participants will have hallux valgus/hallux rigidus surgery using a calf tourniquet which will be removed. There will be a five minute delay before the wound is closed.
  Interventions: Other: Tourniquet release

INTERVENTIONS:
Other: Standard care — Hallux valgus/hallux rigidus surgery with the calf tourniquet remaining in situ until the wound is closed.
  Arms: Standard care
Other: Tourniquet release — Hallux valgus/hallux rigidus surgery with the calf tourniquet released five minutes before the wound is closed.
  Arms: Tourniquet release

SUMMARY:
Patients listed for hallux valgus/hallux rigidus correction surgery will be randomised to one of two treatment groups. Group 1 (standard care) will have the calf tourniquet released after wound closure. Group 2 will have the tourniquet removed five minutes before wound closure. Participants will have the volume of their operated foot measured pre-operatively and post-operatively at six weeks and three months.

DETAILED DESCRIPTION:
Pneumatic tourniquets provide the benefits of better visualisation and decreased blood loss, but can also cause metabolic changes due to ischemia and compressive damage due to pressure. Surveys of foot and ankle surgeons demonstrates prevalent use of tourniquets in their clinical practice, with various patterns of use differing amongst the surgeons.

Bunion surgery is one of the most common surgical procedures in foot surgery. It involves correcting the hallux valgus deformity through a combination of various osteotomy, fusion, or soft tissue procedures. Swelling after any surgery is common, but particularly so after foot surgery as gravity causes fluid to collect in the foot. With regards to recovery after surgery, patients are advised to expect to be off work for between 6-8 weeks for a sedentary occupation, and between 12-14 weeks for heavy work. Although patients have low pain levels, the foot remains swollen for an average of 3-6 months after surgery. It is usually the swelling that prevents patients from getting in to normal footwear to be able to return to work sooner.

Bunion surgery is usually performed under a calf-tourniquet to create a bloodless surgical field and ensure less surgical bleeding, thereby reducing surgical time. However, use of tourniquets can lead to more swelling, increased post-operative pain and challenges in rehabilitation - all of which may affect recovery after bunion surgery. Prolonged duration of tourniquet use has been shown to cause post-operative wound healing complications, potentially attributable to local inflammation and tissue hypoxia. It is known from the studies for knee replacement surgery that tourniquet use can lead to decreased range of motion after surgery in early stage.

This study will be a randomised controlled trial with two study groups. The control group will have surgery with the tourniquet remaining in situ until the wound is closed. The intervention group will have the tourniquet released after surgery, but closure will be delayed by five minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients having hallux valgus or hallux rigidus
* Able to give informed consent
* Able to return for follow-up

Exclusion Criteria:

* Patients with symptomatic peripheral vascular disease
* Patients with known peripheral oedema from any cause
* Patients who will also require lesser toe correction as part of the procedure
* Active smokers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-08-23 (Actual); Primary Completion 2021-08-26 (Estimated); Study Completion 2021-11-25 (Estimated)

PRIMARY OUTCOMES:
Foot volume | 3 months post-operatively
  The volume of the operated foot measured by water displacement (in millilitres).

SECONDARY OUTCOMES:
MOxFQ score | 3 months post-operatively
  Manchester-Oxford Foot Questionnaire score (0-100, 100 being the most severe)
Foot pain assessed using a dolometer | 3 months post-operatively
  Foot pain measured on a visual analogue scale (0-10, 0 being no pain & 10 being worst pain imaginable).
Return to work | 3 months post-operatively
  Time after surgery the participant returned to work (reported in weeks since surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Kalpesh Shah, M.D., Principal Investigator — Gloden Jubilee National Hospital
Locations (1):
- Golden Jubilee National Hospital, Clydebank, West Dunbartonshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No data will be shared